CLINICAL TRIAL: NCT06246175
Title: A Multi-center, Single-dose, Open-label, Parallel Design, Pharmacokinetics Study of HRS9531injection in Healthy Subjects and Subjects With Impaired Renal Function
Brief Title: A Study of HRS9531 in Participants With Impaired Kidney Function and Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-105
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a single-dose, parallel design trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A group (Healthy Control) (Experimental)
  Interventions: Drug: HRS9531
- B group (Mild Renal Impairment) (Experimental)
  Interventions: Drug: HRS9531
- C group (Moderate Renal Impairment) (Experimental)
  Interventions: Drug: HRS9531
- D group (Severe Renal Impairment) (Experimental)
  Interventions: Drug: HRS9531

INTERVENTIONS:
Drug: HRS9531 — Receive a single dose of HRS9531 injection

SUMMARY:
The purpose of this study is to assess how fast HRS9531 gets into the blood stream and how long it takes the body to remove it in participants with impaired kidney function compared to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, be able and willing to provide a written informed consent;
2. Age 18-65 years on the date of signing informed consent (inclusive);
3. Body mass index (BMI) within the range of 19.0-40.0 kg/m2 (inclusive);
4. Renal function, assessed by estimated glomerular filtration rate at screening (eGFR):

   1. Normal renal function: 90-129 mL/min (inclusive);
   2. Mild impairment: 60-89 mL/min (inclusive);
   3. Moderate impairment: 30-59 mL/min (inclusive);
   4. Severe impairment: 15-29 mL/min (inclusive);
5. Females of childbearing potential should have negative baseline blood pregnancy test, and must use highly effective contraception from signing the informed consent form to 2 months after the last dose of trial drug; Male subjects must agree to either remain abstinent or use highly effective contraceptive measures during the trial and 2 months after last dose of the trial drug, or have been surgically sterilized;
6. Stable renal function, assessed by two eGFR during screening (apart at least 3 days);
7. Diagnosed as stable, chronic renal disease for at least 3 months.

Exclusion Criteria:

1. Have any GI disease which impacts gastric emptying (eg, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy);
2. Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2; Have a history or presence of pancreatitis;
3. Had a severe trauma or major surgery within 6 months prior to screening, planned to undergo surgery during the trial period;
4. Participants in clinical trials of any drug or medical device in the 3 months prior to screening;
5. Blood donation history or blood loss ≥400 mL within 3 month or ≥200 mL within 1 month before screening, or received blood transfusion within 3 months;
6. Allergic constitution includes severe drug allergy or history of drug allergy;
7. Hepatitis B surface antigen (HBsAg), HIV antibody detection, hepatitis C virus antibody (HCVAb), treponema pallidum specific antibody detection, positive;
8. Regularly use known drugs of abuse and/or show positive findings on urinary drug screen that are not otherwise explained by permitted concomitant medications;
9. Have an average weekly alcohol intake that exceeds 14 units per week or average daily cigarettes consumption exceeds 5 per day, and are unwilling to stop alcohol or cigarettes consumption 24 hours prior to dosing until discharge from the study or completion of all study procedures (1 unit =12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits);
10. History use of GLP-1R（glucagon-like peptide-1 receptor） agonist, GLP-1R/GCGR（glucagon receptor）agonist, GIPR（glucose-dependent insulinotropic polypeptide receptor/GLP-1R agonist or GIPR/GLP-1R/GCGR agonist within 2 months prior to screening;
11. Breast-feeding women;
12. The use of alcohol- or caffeine-containing foods or beverages within 72 hours prior to Check-in (Day -1), unless deemed acceptable by the investigator;
13. History of Vasovagal Syncope; Do not have venous access sufficient to allow blood sampling as per the protocol；
14. The need to follow a special diet and unable to follow the diet requirement of protocol;
15. The investigator considers that the subject has any other factors that would make it inappropriate to participate in this study
16. Healthy Participants:

    1. Systolic blood pressure <90 mmHg or ≥140 mmHg; Diastolic blood pressure <50 mmHg 或≥90 mmHg; Heart Rate < 50 beats/min or >100 beats/min;
    2. Have a significant history or presence of cardiovascular (eg, myocardial infarction, cerebrovascular accident, etc. within the past 6 months), respiratory, hepatic, renal, GI, endocrine (except T2DM), haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data;
    3. Use of medications determined to be unsuitable by the investigator (including over-the-counter medication, prescription medication and herbal preparations) within the 14 days prior to screening;
    4. Have clinical laboratory test results outside normal reference range for the population or investigator site and judged to be clinically significant by the investigator;
17. Participants with Renal Impairment：

    1. Systolic blood pressure <90 mmHg or≥160 mmHg; Diastolic blood pressure <50 mmHg 或 ≥100 mmHg; Heart Rate < 50 beats/min or >100 beats/min;
    2. Have a significant history or presence of cardiovascular (eg, myocardial infarction, cerebrovascular accident, decompensated heart failure (NYHA classification III or IV), etc. within the past 6 months), respiratory, hepatic, renal (obstructive urinary tract disease, except CKD), GI, endocrine (except T2DM), haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data;
    3. History of Kidney Transplant;
    4. Subjects started new over-the-counter or prescription medications (eg, antihypertensive agents, aspirin, lipid-lowering agents) for treatment of concurrent medical conditions or on their treatment regimen for less than 1 month;
    5. Have following clinically relevant abnormal laboratory test results:

       * Hemoglobin <85 grams per liter (g/L);
       * Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3× the upper limit of normal (ULN) or total bilirubin (TBL) >1.5× ULN;
       * Serum triglyceride > 5.64 mmol/L（500 mg/dl）;
       * Clinical relevant elevation in serum amylase or lipase；
       * QTcF > 450 msec;
       * Other abnormal lab results, as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve (AUC) of HRS9531 From Time Zero to Tlast (AUC0-t) | Start of Treatment up to Day 29
Maximum Concentration of HRS9531 (Cmax) | Start of Treatment up to Day 29
Area Under the Concentration Versus Time Curve (AUC) of HRS9531 From Time Zero to Infinity (AUC0-inf) | Start of Treatment up to Day 29

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Start of Treatment up to Day 29
Apparent terminal half-life (t1/2) | Start of Treatment up to Day 29
Apparent clearance (CL/F) | Start of Treatment up to Day 29
Apparent volume of distribution (Vz/F) | Start of Treatment up to Day 29
Incidence and severity of adverse events | Screening period up to Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided